CLINICAL TRIAL: NCT03183843
Title: The Use of Dabigatran Etexilate in Patients With Atrial Fibrillation After Mitral Valve Prosthetic Replacement
Brief Title: Dabigatran in Patients With Atrial Fibrillation and Mitral Biological Prostheses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Sergey Mamchur, Head of Department of Cardiovascular Disorders Diagnosis, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0546-2015-0011
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Mitral Valve Stenosis and Insufficiency; Atrial Fibrillation
Keywords: Atrial Fibrillation; Mitral Valve Stenosis; Mitral Valve Insufficiency; Dabigatran; Biological Prosthesis; Mitral Valve Replacement; Cox-Maze Procedure
MeSH Terms: conditions — Mitral Valve Stenosis; Atrial Fibrillation; Mitral Valve Insufficiency | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dabigatran (Active Comparator): Dabigatran etexilate 150 mg by mouth every 12 hours for a year
  Interventions: Drug: Dabigatran Etexilate
- Warfarin (Active Comparator): Warfarin by mouth every 24 hours in a dose providing international normalized ratio (INR) 2.5-3.5 for a year
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran Etexilate — Dabigatran Etexilate 150 mg capsules for oral administration twice a day
  Other Names: Pradaxa
  Arms: Dabigatran
Drug: Warfarin — Warfarin 2.5 mg tablets for oral administration once a day
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
The efficacy and safety of anticoagulation therapy using dabigatran in comparison with warfarin will be evaluated in patients with atrial fibrillation after mitral valve prosthetic replacement concomitant with Cox-Maze procedure.

DETAILED DESCRIPTION:
Patients with prosthetic mitral valves need a long-term anticoagulation therapy. After mitral valve replacement using mechanical prostheses warfarin is administrated during the whole life. Biological prostheses allows do discontinue anticoagulation 3 months after surgery in the absence of other risk factors of thrombosis especially atrial fibrillation. The common approach to patients with mitral valve disease and atrial fibrillation is mitral valve prosthetic replacement concomitant to Cox-Maze procedure. This allows to maintain sinus rhythm in 65-80% of patients. In the study the safety and efficacy of dabigatran in comparison with warfarin will be evaluated after the mitral valve surgery and Cox-Maze procedure.

ELIGIBILITY:
Inclusion Criteria:

* mitral valve disease;
* atrial fibrillation;
* mitral valve prosthetic replacement with concomitant Cox-Maze Procedure;
* 18-75 years of age;
* signed informed consent form.

Exclusion Criteria:

* mechanical valve replacement;
* repeated mitral valve surgery;
* coronary artery hemodynamically significant stenoses;
* ventricular arrhythmias;
* creatinine clearance <50 ml/min;
* HAS-BLED score >3;
* previous stroke or transient ischemic attack;
* liver diseases;
* neoplasia;
* pregnancy;
* simultaneous antiplatelet therapy;
* allergic reactions on Dabigatran or Warfarin;
* cognitive disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Thrombosis | 1 year
  Thrombosis of prosthetic valve, transient ischemic attack, stroke, myocardial infarction, pulmonary and systemic thromboembolic events

SECONDARY OUTCOMES:
Major Bleeding | 1 year
  Massive symptomatic intracranial, intraocular, retroperitoneal, intraarticular, pericardial bleeding or intramuscular bleeding associated with compressive syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yevgeny V Grigoriev, M.D., Ph.D., Study Chair — Research Institute for Complex Problems of Cardiovascular Diseases
Locations (1):
- Research Institute for Complex Problems of Cardiovascular Diseases, Kemerovo, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadlapati A, Groh C, Malaisrie SC, Gajjar M, Kruse J, Meyers S, Passman R. Efficacy and safety of novel oral anticoagulants in patients with bioprosthetic valves. Clin Res Cardiol. 2016 Mar;105(3):268-72. doi: 10.1007/s00392-015-0919-z. Epub 2015 Sep 18. PMID 26384981
- [Background] Sun JC, Davidson MJ, Lamy A, Eikelboom JW. Antithrombotic management of patients with prosthetic heart valves: current evidence and future trends. Lancet. 2009 Aug 15;374(9689):565-76. doi: 10.1016/S0140-6736(09)60780-7. PMID 19683642